CLINICAL TRIAL: NCT02865135
Title: A Phase Ib/II Trial To Test The Safety And Efficacy Of Vaccination With HPV16-E711-19 Nanomer For The Treatment Of Incurable HPV 16-Related Oropharyngeal, Cervical And Anal Cancer In HLA-A*02 Positive Patients
Brief Title: Trial To Test Safety And Efficacy Of Vaccination For Incurable HPV 16-Related Oropharyngeal, Cervical And Anal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Principal Investigator, Kartik Sehgal, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-578
Record Dates: First submitted 2016-07-14; First posted 2016-08-12 (Estimated); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Cancer of Head and Neck; Cancer of Cervix; Cancer of Anus
Keywords: HPV Related Head and Neck; Cervical; Anal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Uterine Cervical Neoplasms; Anus Neoplasms | interventions — Papillomavirus Vaccines; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DPX-E7 + Cyclophosphamide [Phase Ib Cohort] (Experimental): Participants received: 1) 50 mg twice per day of cyclophosphamide orally 7 days before the vaccination, continuing for 7 days on and then 7 days off, throughout the treatment period; 2) two 0.25 mL priming doses of DPX-E7 3 weeks apart, followed by 0.1 mL booster dose every 8 weeks until clinical progression.
  Interventions: Drug: DPX-E7 vaccine; Drug: Cyclophosphamide
- DPX-E7 + Cyclophosphamide [Phase II Cohort 1] (Experimental): Participants were enrolled before amendment 10. Participants received: 1) 50 mg twice per day of cyclophosphamide orally 7 days before the vaccination, continuing for 7 days on and then 7 days off, throughout the treatment period; 2) two 0.25 mL priming doses of DPX-E7 3 weeks apart, followed by 0.1 mL booster dose every 8 weeks until clinical progression.
  Interventions: Drug: DPX-E7 vaccine; Drug: Cyclophosphamide
- DPX-E7 [Phase II Cohort 2] (Experimental): Participants were enrolled after amendment 10. Participants received two 0.50 mL priming doses of DPX-E7 3 weeks apart, followed by 0.2 mL booster dose every 8 weeks until clinical progression.
  Interventions: Drug: DPX-E7 vaccine

INTERVENTIONS:
Drug: DPX-E7 vaccine — Therapeutic vaccine for the treatment of incurable HPV16-related oropharyngeal, cervical and anal cancer in HLA-A*02 positive patients.
  Other Names: HPV vaccine
Drug: Cyclophosphamide — Cyclophosphamide is a medication primarily used in the management and treatment of neoplasms, including multiple myeloma, sarcoma, and breast cancer. Cyclophosphamide is a nitrogen mustard that exerts its anti-neoplastic effects through alkylation.
  Other Names: Cytoxan
  Arms: DPX-E7 + Cyclophosphamide [Phase II Cohort 1]; DPX-E7 + Cyclophosphamide [Phase Ib Cohort]

SUMMARY:
This research study is studying a therapeutic vaccine, named DPX-E7, as a possible treatment for Human Papilloma Virus or HPV related head and neck, cervical or anal cancer (positive for HLA-A*02).

DETAILED DESCRIPTION:
This is a phase Ib/II clinical trial. DPX-E7 is a therapeutic vaccine, intended to treat HPV-related head and neck, cervical or anal cancer. DPX-E7 is an investigational vaccine and the FDA (the U.S. Food and Drug Administration) has not approved DPX-E7 vaccine as a treatment for any disease.

DPX-E7 is being tested in humans for the first time. DPX-E7 is a kind of immunotherapy that will make the immune system to elicit an anti-tumor response by generating CD8+ T-cells. CD8+ T-cells play a very important role in fighting against viral infections

ELIGIBILITY:
Inclusion Criteria:

* Each patient must be positive for HLA-A*02 and meet all of the following inclusion criteria to be enrolled in the study:
* Histologically or cytologically proven HPVOC or cervical cancer or anal cancer, based on expression of HPV type16 in immunohistochemistry and/or HPV 16 DNA analysis by ISH of tumor tissue from the primary or metastatic lesions.
* Incurable HPVOC, as defined by:

  * Relapsed or progressive disease at the primary site and/or regional lymph nodes after initial treatment (e.g. Surgery, radiotherapy or chemoradiotherapy) with no potentially curative option (i.e. surgery or radiation); OR
  * Distant metastasis
* Incurable cervical or anal cancer, as defined by:

  * Relapsed or progressive disease at the primary site and/or regional lymph nodes after initial treatment (e.g. systemic chemotherapy) with no potentially curative option (i.e. surgery or chemoradiotherapy). Chemotherapy administered in conjunction with primary radiation as a radiosensitizer will not be counted as a systemic chemotherapy regimen; OR
  * Distant metastasis refractory to initial treatment (at least one prior chemotherapeutic regimen which can include a single chemotherapeutic, a combination of chemotherapeutics, or biologic drugs such as bevacizumab).
* Accessible tumors for sequential biopsies Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.03) to grade 1 or better (except for < grade 2 neuropathy, alopecia, xerostomia, dysphagia, or mucositis);
* Age ≥ 18 years;
* Measurable disease, according to modified RECIST 1.1 and irRECIST (Appendix B & C);
* Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 2 (Appendix A)
* Adequate bone marrow, liver and renal function, defined by:

  * Hemoglobin ≥ 10 g/dL;
  * Absolute neutrophil count (ANC) ≥ 1000/μL;
  * Absolute lymphocyte count ≥ 400/μL;
  * Platelet count ≥ 100,000/μL;
  * ALT and AST ≤ 2.5 X upper limit of normal (ULN);
  * Total bilirubin ≤ 1.5 X ULN; and
  * Serum creatinine ≤ 1.5 X ULN;
* Women of child-bearing potential (WOCBP) must be willing to use acceptable means of birth control;
* Men who could potentially father a child must also use birth control
* Signed informed consent

Exclusion Criteria:

* Radiotherapy for primary HPVOC within 8 weeks, or radiotherapy for any other reason within 3 weeks prior to the first dose of trial treatment;
* Chemotherapy within 3 weeks prior to the first dose of trial treatment;Other cancer in the past 5 years, except for carcinoma in situ of the cervix or bladder, or non-melanomatous skin cancer;
* Inaccessible tumor or lack of consent for sequential biopsies
* Uncontrolled central nervous system (CNS) metastases (i.e. known CNS lesions that are radiographically unstable, symptomatic and/or requiring escalating doses of corticosteroids);
* Active hepatitis, known HIV, or other condition that requires immunosuppressive therapy, including current use of high dose systemic corticosteroids;
* Autoimmune disease, such as systemic lupus erythematosis or rheumatoid arthritis, that is active and requires current immunosuppressive therapy;
* Active uncontrolled serious infection;
* WOCBP who have a positive β-hCG test or are breastfeeding.
* Acute or chronic skin disorders that would interfere with subcutaneous injection of the vaccine or subsequent assessment of potential skin reactions;
* Allergies to any vaccine, that after discussion with Immunovaccine, are serious enough to warrant exclusion from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Seghal, MD, Principal Investigator — Dana-Farber Cancer Institute, Boston, MA02215
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from 3/30/17 until 9/10/19.
Period: Overall Study
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] | DPX-E7 [Phase II Cohort 2]
Started | 6 | 3 | 2
Evaluable for T Cell Analysis | 6 | 3 | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 3 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Progression | 6 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] | DPX-E7 [Phase II Cohort 2] | Total
Number analyzed (Participants) | 6 | 3 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (11.9) | 54.1 (9.29) | 69.5 (1.76) | 56.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 4 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 3 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group Performance Score (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS0: Fully active, able to carry on all pre-disease performance without restriction ECOG PS1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG PS2: Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about more than 50% of waking hours.
  Participants
    ECOG PS0 | 3 | 1 | 1 | 5
    ECOG PS1 | 2 | 2 | 1 | 5
    ECOG PS2 | 1 | 0 | 0 | 1
Site of Disease [Count of Participants; unit: Participants]
  Anal | 1 | 1 | 0 | 2
  Cervical | 5 | 1 | 2 | 8
  Oropharyngeal | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) [Phase 1b]
Description: A DLT was defined as any grade 3 or greater adverse event at least possibly related to the study agent including injection site reactions; or grade 2 or greater allergic reactions which occur in a subject prior to day 50, will trigger DLT. In addition, to be considered as DLT, the adverse event must be considered at least possibly related to study treatment. Grade 3 or greater abnormal lab values lasting <= 72 hours might be excluded as DLTs if there are no accompanying clinical signs and symptoms per investigator's discretion.
Time Frame: Patients were followed for 50 days.
Measure: Count of Participants; unit: Participants
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort]
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Grade 1-2 Treatment-Related AE Rate
Description: The proportion of participants who experienced grade 1-2 treatment-related adverse events based on the Common Toxicity Criteria for Adverse Events Version 4.0 (CTCAEv4) as reported on case report forms.
Time Frame: The median follow up was 2.92 months (range 1.25 - 5.88months).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] | DPX-E7 [Phase II Cohort 2]
Number analyzed (Participants) | 6 | 3 | 2
proportion of participants | 0.66 [0.22 to 0.96] | 1 [0.01 to 1] | 1 [0 to 1]

3. Primary Outcome: Changes in CD8+ T Cells in Peripheral Blood and Tumor Tissue
Description: 'Responders' will be defined as patients with at least a two-fold increase in the number of CD 8+ T cells (dextramer, ELISpot or both methods) in the peripheral blood and tissue at the final analysis.
Time Frame: Patients were followed 22 days.
Population: Data were not collected for participants who registered after amendment 10.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] | DPX-E7 [Phase II Cohort 2]
Number analyzed (Participants) | 6 | 3 | 0
percentage of participants
  Responders | 16.7 [0.6 to 64.1] | 0 [0 to 70.8] |
  Non-responder | 83.3 [35.9 to 99.6] | 100 [29.2 to 100] |

4. Secondary Outcome: Best Overall Response
Description: Best Overall Response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started) based on modified RECIST 1.1 and irRECIST. Per irRECIST, CR was defined as disappearance of all lesions in two consecutive observations not less than four weeks apart; PR was defined as greater than or equal to 50% decrease in tumor burden compared with baseline in two observations at least four weeks apart.
Time Frame: The median follow up was 2.92 months (range 1.25 - 5.88months).
Measure: Count of Participants; unit: Participants
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] | DPX-E7 [Phase II Cohort 2]
Number analyzed (Participants) | 6 | 3 | 2
Participants
  SD | 2 | 1 | 0
  PD | 4 | 1 | 2
  Unevaluable | 0 | 1 | 0

5. Secondary Outcome: Median Overall Survival
Description: Overall survival based on the Kaplan-Meier method is defined as the time the start of treatment to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.
Time Frame: The median follow up was 4.8 months (range 1.6 - 14.9 months).
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] | DPX-E7 [Phase II Cohort 2]
Number analyzed (Participants) | 6 | 3 | 2
Months | 16.5 [1.8 to 16.5] | 4.8 [3.7 to 5.9] | NA [NA to NA] — Limited number of participants died during the time of observation.

6. Secondary Outcome: Median Progression-Free Survival
Description: PFS is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anticancer therapy. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study or the appearance of one or more new lesions. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: The median follow up was 4.8 months (range 1.6 - 14.9 months).
Population: The analysis dataset is comprised of all enrolled participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] | DPX-E7 [Phase II Cohort 2]
Number analyzed (Participants) | 6 | 3 | 2
Months | 2.9 [1.2 to 4.8] | 3.3 [2.8 to 5.9] | 1.4 [1.2 to 1.6]

7. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study. Participants alive without PD were censored at the earliest of the date of the last disease evaluation. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study or the appearance of one or more new lesions. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: The median follow up was 4.8 months (range 1.6 - 14.9 months).
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] | DPX-E7 [Phase II Cohort 2]
Number analyzed (Participants) | 6 | 3 | 2
Months | 2.9 [1.2 to 4.8] | 3.3 [2.8 to 5.9] | 1.4 [1.2 to 1.6]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time that participants signed consent and 30 days post treatment-end. Participants received a median (range) treatment duration in months 2.92 (1.25 - 5.88). Deaths were monitored until 14.9 months.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Per the source vocabulary (CTCAEv4.0) there is a category "Other, specify" for each system organ class. No further data is available to specify classification beyond this general term.
Arm/Group | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] | DPX-E7 [Phase II Cohort 2]
All-Cause Mortality (participants affected / at risk) | 3/6 | 2/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/3 | 1/2
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] (N=6) | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] (N=3) | DPX-E7 [Phase II Cohort 2] (N=2)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Death NOS (General disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DPX-E7 + Cyclophosphamide [Phase Ib Cohort] (N=6) | DPX-E7 + Cyclophosphamide [Phase II Cohort 1] (N=3) | DPX-E7 [Phase II Cohort 2] (N=2)
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 4 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 6 | 2 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Edema face (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 6 | 2 | 1
Fever (General disorders) | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Cholesterol high (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0
Genital edema (Reproductive system and breast disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 1 | 0

LIMITATIONS AND CAVEATS:
Week accrual leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT02865135/Prot_SAP_000.pdf